CLINICAL TRIAL: NCT01897090
Title: The Relationship of a "Crohn's Disease Diet" in Reducing Symptoms of Crohn's Disease, Improving Quality of Life, and Decreasing Related Health Care Costs.
Brief Title: A Crohn's Disease Diet to Reduce Symptoms of Crohn's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Johns Hopkins University (Other)
Collaborators: The Broad Foundation (Other)
Responsible Party: Principal Investigator, Gerard E. Mullin, Associate Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00042692
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Crohn's Disease
Keywords: Elimination Diet; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Elimination Diets; Nutrition Policy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elimination Diet (Experimental): thirty (30) patients will be on the "Crohn's Disease Diet" (primarily an "anti-inflammatory diet that is an elimination diet - gluten-free, casein-free based with limited carbohydrate)
  Interventions: Other: Elimination Diet
- Dietary Guidelines for Americans (Active Comparator): The DASH eating plan is based on 1,600, 2,000, 2,600 and 3,100 calories.
  Interventions: Other: Dietary Guidelines for Americans

INTERVENTIONS:
Other: Elimination Diet
  Arms: Elimination Diet
Other: Dietary Guidelines for Americans
  Arms: Dietary Guidelines for Americans

SUMMARY:
A 16-week randomized, pilot study to determine if an elimination diet reduces symptoms of Crohn's disease. Sixty (60) adult patients (18-75 yrs) with a mild or moderate Crohn's Disease Activity Index (CDAI) of 150-450, will be recruited through the GI practices at Johns Hopkins University. Patients agree not to be on any other major treatments, with the exception of consistent/stable doses of 5-aminosalicylate (ASA) drugs/other medications during the course of the study and will obtain their physician's permission.They will be divided into a treatment and standard diet group: thirty (30) patients will be on the "Crohn's Disease Diet" (primarily an "anti-inflammatory diet that is an elimination diet - gluten-free, casein-free based with limited carbohydrate) and thirty (30) patients will be given the Dietary Guideline recommendations and similar dietary counseling attention. To assess the clinical efficacy and tolerance of the trial population, patients will be monitored by two office visits (at 0 and 12 weeks) by visits with the Clinical Research Unit (CRU) registered dietitians (RDs) at 0, 6, 12, and 16 weeks (4 weeks after the end of the study) for blood and dietary data collection. Clinical endpoints will be Crohn's disease Activity Index (CDAI) scores (remission < 150; mild = 150-220; moderate = 220-450; severe = 450+), C-Reactive Protein (CRP) values (0-0.8 mg/L), sedimentation rate /(male: 15-20 mm/hr, female: 20-30 mm/hr)/, possibly interleukin-6(/normal value: <10pg/ml)/, Overall Quality of Life (QOL) through the Inflammatory Bowel Disease Questionnaire (IBDQ), Dudley IBD Symptom Questionnaire (DISQ) surveys, and Brown's Gastrointestinal Quality of Life (QOL) Questionnaire, and health care costs measured by a health care cost questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age with any gender.
* Between 150-220 or moderate Crohn's Disease with a CDAI between 220-450.
* Not a smoker.
* No current signs or symptoms of severe, progressive or uncontrolled renal, gastroenterological, hepatic, hematological, endocrine, pulmonary, cardiac, neurological or cerebral disease.
* Understand and be able to adhere to the dosing and visit schedules; and agree to record symptom severity scores, any medications or dietary supplements, and adverse events accurately and consistently in a daily diary.
* Agree during the study to use only the designated therapy, however, patients will qualify for the study if they are on a 3-month stable dose of 5-ASA or immunomodulators and there is a limited change in medication dosage no minimize biasing the results.
* Agree that you have not previously followed diets where you have eliminated an allergen, lactose, gluten or major food group for the purpose of reducing Crohn's disease symptoms within the last year.
* Agree not to use any oral medications, dietary supplements, herbal treatments, diet therapies within three weeks of the onset of the trial or during the study. During the study agree to use only the designated therapy, however, patients will qualify for the study if they are on a 3-month stable dose of 5-aminosalicylic acid (ASA) or immunomodulators and there is a limited change in medication dosage no minimize biasing the results.
* Willing to follow the diet during the study and to weigh themselves weekly.

Exclusion Criteria:

* Have extensive colonic, ileal or ileocolonic resection, ileostomies or colostomies with ileal pouch.
* Experiencing severe weight loss (if % of weight change within 1 week >2% or 1 month >5% or 3 months >7.5% or 6 months > 10%) or severely malnourished (if < 74% of usual body weight).
* Pregnant, lactating woman or desire to become pregnant during the study. [ ] [ ] Patients receiving prescribed oral nutrition and/or intravenous nutrition.
* Presence of alcohol, drug abuse, or smoking (cigarette or other).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
CDAI score | 16 weeks
  Clinical endpoints will be Crohn's disease Activity Index (CDAI) scores (remission < 150; mild = 150-220; moderate = 220-450; severe = 450+),

SECONDARY OUTCOMES:
CRP | 16 WEEKS
  C-Reactive Protein (CRP) values (0-0.8 mg/L)
sed rate | 16 weeks
  sedimentation rate (male: 15-20 mm/hr, female: 20-30 mm/hr)
Quality of Life | 16 weeks
  Score on short inflammatory bowel disease questionniare (SIBDQ) and Brown's GI Quality of Life measure
Symptom improvement | 16 weeks
  Score of DISQ

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Brown AC, Roy M. Does evidence exist to include dietary therapy in the treatment of Crohn's disease? Expert Rev Gastroenterol Hepatol. 2010 Apr;4(2):191-215. doi: 10.1586/egh.10.11. PMID 20350266
- [Background] Brown AC, Rampertab SD, Mullin GE. Existing dietary guidelines for Crohn's disease and ulcerative colitis. Expert Rev Gastroenterol Hepatol. 2011 Jun;5(3):411-25. doi: 10.1586/egh.11.29. PMID 21651358
- See also: The Broad Foundation — http://www.broadfoundation.org/